CLINICAL TRIAL: NCT01066637
Title: Imaging iNOS Activity Using [18F] (+/-) NOS With Positron Emission Tomography (PET) in Cellular Inflammation.
Brief Title: iNOS With Positron Emission Tomography (PET) in Cellular Inflammation.
Acronym: F-NOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0986; 201106273 (Registry Identifier: myIRB HRPO)
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Patients With Post Orthotopic Heart Transplantation Status
Keywords: Heart transplant patients
MeSH Terms: interventions — Fluorine-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dosimetry Group (Experimental): To determine its potential for use in humans, we measured 18F-NOS myocardial activity in patients after orthotopic heart transplantation (OHT) (3 women and 9 men) and normal healthy volunteers (2 women and 2 men), and correlated it with pathologic allograft rejection, tissue iNOS levels, and calculated human radiation dosimetry.
  Interventions: Drug: [18F](+/-)NOS
- Kinetic Analysis Group (Experimental): Measurement of myocardial levels of enzyme nitric oxide synthase(iNOS) using PET and 18F-NOS in post heart transplant patients (5 women and 5 men) undergoing endomyocardial biopsy as part of their normal post-transplant evaluation. Kinetic data of the tracer will be compared with the heart tissue measurements of iNOS measured by immunohistochemistry.
  Interventions: Drug: [18F](+/-)NOS

INTERVENTIONS:
Drug: [18F](+/-)NOS — Injection of radiotracer [18F](+/-)NOS for PET imaging and kinetic data analysis
  Other Names: 6-(1/2)(2-18F-fluoropropyl)-4-methylpyridin-2-amine

SUMMARY:
The primary purpose of this study is to measure the level of an enzyme in a patient's heart called inducible nitric oxide synthase(iNOS) using Positron Emission Tomography (PET) imaging with a radioactive tracer called 18F-NOS. These PET results will be compared to tissue results obtained during routine endomyocardial heart biopsy. The enzyme iNOS produces nitric oxide in inflammatory diseases such as acute heart transplant rejection, diabetes, Alzheimer's and cancer. Thus, PET with the radioactive tracer 18F-NOS may be a useful tool for detecting the early stages of these diseases. The safety of 18F-NOS during the study will also be assessed. All PET imaging will be performed with a CTI/Siemens Biograph 40 PET/CT scanner. Protocol was revised to add new imaging modality, Biograph mMR PET-MR scanner in order to investigate new hardware and software in order to optimize scanning procedures in order to refine image quality so that we can apply the findings to future standard clinical scans and research imaging studies. Ten additional status-post OHT patients who are scheduled for standard of care endomyocardial biopsy for allograft rejection surveillance will undergo PET/MR imaging with [18F](+/-)NOS.

DETAILED DESCRIPTION:
Nitric oxide (NO) is an important and unique mediator of a variety of physiological and pathological processes. NO is generated from the oxidation of L-arginine to L-citrulline in a two-step process by nitric oxide synthase (NOS) enzymes. In the NOS family, there are two constitutive isozymes of NOS, neuronal NOS (nNOS) and endothelial NOS (eNOS), and one inducible isozyme (iNOS). The three isozymes of NOS are expressed in different tissues to generate NO for specific physiological roles. nNOS generates NO as a neurotransmitter and neuromodulator, mainly in brain and peripheral nerve cells; eNOS regulates blood pressure, and blood flow primarily in vascular endothelial cells. The induction of iNOS occurs by various inflammatory stimuli (e.g., endotoxin) in activated macrophages and other types of cells and plays a crucial role in the host defense and the inflammatory processes.

Normally, the basal level of NO in all parts of the body is very low, mainly due to the constitutive nNOS and eNOS. In contrast, once expressed, iNOS can continue to generate NO in large amounts (up to μM concentrations) for a prolonged period of time. Studies have shown that production of NO by iNOS is implicated in a variety of acute and chronic inflammatory diseases (e.g., sepsis, septic shock, organ transplant rejection, vascular dysfunction in diabetes, asthma, arthritis, multiple sclerosis, and inflammatory diseases of the gut). iNOS activity has also been found in many tumors. Because of the central role of iNOS in NO-related diseases, numerous efforts have been made to develop iNOS inhibitors as pharmaceuticals ranging from the nonselective L-arginine analogues to the selective inhibitors reported recently. Some inhibitors of iNOS have shown promising results in animal models of sepsis, lung inflammation, arthritis, and autoimmune diabetes. Therefore, the development of a radiolabeled iNOS inhibitor for probing iNOS expression in vivo using noninvasive positron emission tomography (PET) imaging will be of tremendous value to the study and treatment of NO-related diseases.

Acute allograft rejection is the major contributor to mortality in patients receiving orthotopic heart transplantation (OHT). Specifically, iNOS has been thought to be the main NOS involved in producing NO that is active in acute cardiac allograft rejection. Up-regulation of iNOS occurs in macrophage cellular infiltrates and later within the graft parenchymal cells. In human cardiac transplantation a positive correlation has shown between iNOS expression and left ventricular contractile dysfunction measured by echocardiography and Doppler techniques. We have recently developed a novel PET radiotracer, [18F](+/-)NOS, designed to measure cellular iNOS activity. This study evaluates the feasibility of the method in OHT patients undergoing surveillance endomyocardial biopsy as part of their normal post-transplant evaluation for potential allograft rejection. More specifically, it will compare the myocardial kinetics of this radiotracer measured by PET with tissue measurements of iNOS measured by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

1. The OHT patients will be undergoing surveillance endomyocardial biopsy and will Patients 21 years of age or older of either sex, who are status-post OHT and normal healthy volunteers (2 women and 2 men) will be enrolled.be on standard immunosuppressive therapy and anti-hyperlipidemic, anti-hypertensive and anti-diabetic therapies as needed. "Healthy volunteer" is someone who has volunteered to be imaged and who, based on physical exam and baseline electrocardiogram, has no evidence of cardiovascular disease, is not on medication, such as steroids, that will interfere with the accuracy of measuring [18F](+/-)NOS activity and is not under the care of a physician for any active medical conditions.
2. Able to give informed consent.
3. Not currently pregnant or nursing: Female subjects must be either: surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post menopausal (cessation of menses for more than 1 year), or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of [18F](+/-)NOS) is negative.

Exclusion Criteria:

1. Patients with an unstable cardiovascular (e.g., severe rejection) or other clinical condition (e.g., active severe infection) that in the opinion of the Principal Investigator or designee or Dr. Ewald precludes participation in the study.
2. Unable to tolerate 60-90 mins of PET imaging or is claustrophobic.
3. Normal volunteers with evidence of cardiovascular disease or other diseases based on clinical evaluation and/or blood laboratory tests, which are judged by the Principal Investigator or designee to interfere with accurate determination of the of [18F](+/-)NOS on such measures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Gropler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marletta MA. Nitric oxide synthase structure and mechanism. J Biol Chem. 1993 Jun 15;268(17):12231-4. No abstract available. PMID 7685338
- [Background] Kaneki M, Shimizu N, Yamada D, Chang K. Nitrosative stress and pathogenesis of insulin resistance. Antioxid Redox Signal. 2007 Mar;9(3):319-29. doi: 10.1089/ars.2006.1464. PMID 17184170
- [Result] Alderton WK, Cooper CE, Knowles RG. Nitric oxide synthases: structure, function and inhibition. Biochem J. 2001 Aug 1;357(Pt 3):593-615. doi: 10.1042/0264-6021:3570593. PMID 11463332
- [Result] Mollace V, Muscoli C, Masini E, Cuzzocrea S, Salvemini D. Modulation of prostaglandin biosynthesis by nitric oxide and nitric oxide donors. Pharmacol Rev. 2005 Jun;57(2):217-52. doi: 10.1124/pr.57.2.1. PMID 15914468

RESULTS

PARTICIPANT FLOW:
Groups:
- Dosimetry Group: To determine its potential for use in humans, we measured 18F-NOS myocardial activity in patients after orthotopic heart transplantation (OHT) (9 women and 9 men) and normal healthy volunteers (2 women and 2 men), and correlated it with pathologic allograft rejection, tissue iNOS levels, and calculated human radiation dosimetry.
  [18F](+/-)NOS: Injection of radiotracer [18F](+/-)NOS for PET imaging and kinetic data analysis
Period: Overall Study
Arm/Group | Dosimetry Group | Kinetic Analysis Group
Started | 16 | 10
Completed | 16 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dosimetry Group-measuring Radioisotope in Blood: To determine its potential for use in humans, we measured the level of 18F-NOS radiopharmaceutical in patients after orthotopic heart transplantation (OHT) (3 women and 9 men) and normal healthy volunteers (2 women and 2 men), and correlated it with pathologic allograft rejection, tissue iNOS levels, and calculated human radiation dosimetry.
  The level of 18-F-NOS was measured at different time points in minutes after injection of the radioisotope: The measurement time points were 0/120 minutes, 30/150 minutes, 60/180 minutes, and 90/210 minutes. The imaging began from mid thigh, to the base of the brain.
- Kinetic Analysis Group-measuring Levels of Nitric Oxide: Measurement of myocardial levels of enzyme nitric oxide synthase(iNOS) using PET and 18F-NOS in post heart transplant patients (5 women and 5 men) undergoing endomyocardial biopsy as part of their normal post-transplant evaluation. Kinetic data of the tracer will be compared with the heart tissue measurements of iNOS measured by immunohistochemistry.
- Total: Total of all reporting groups
Arm/Group | Dosimetry Group-measuring Radioisotope in Blood | Kinetic Analysis Group-measuring Levels of Nitric Oxide | Total
Number analyzed (Participants) | 16 | 10 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 10 | 26
Dosimetry and Kinetics [Count of Participants; unit: Participants] — Dosimetry group unit of measure which measures the level of radioisotopes in blood uses millicures, which is the unit of measurement to measure radioisotopes in blood. A millicure is a unit of radioactivity equal to one thousandth of a cure;3.70 x disintegrations per second.
  Kinetics is the unit of measurement to measure the amount of INOS in the blood. INOS is an enzyme which catalyses the production of nitroc oxide. Population: The PI has left the institution and we no longer have access to this data.

OUTCOME MEASURES:

1. Primary Outcome: To Measure Free Fatty Acid by Imaging Patients With Increased Levels of iNOS Using [18F](+/-)NOS.
Time Frame: 24-72 hours post [18F](+/-)NOS injection
Population: The PI has left the institution and all efforts to locate data have been exhausted. There is no access to study data and it therefore cannot be reported.
Arm/Group | Dosimetry Group | Kinetic Analysis Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Determine Human Dosimetry in Both Normal Adult Healthy Volunteers and Heart Transplant Patients.
Description: All subjects will receive a single intravenous administration of 7 mCi of [18F](+/-)NOS followed by dynamic PET/CT imaging
Time Frame: 24-72 hours post [18F](+/-)NOS injection
Population: as for outcome 1
Arm/Group | Dosimetry Group | Kinetic Analysis Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1-2 days
Arm/Group | Dosimetry Group | Kinetic Analysis Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/10

LIMITATIONS AND CAVEATS:
there were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes